CLINICAL TRIAL: NCT03314246
Title: Development and Implementation of Ramadan "Fasting Algorithm for Singaporeans With Type 2 Diabetes" (FAST): A Prospective Randomized Controlled Intervention Study
Brief Title: Development and Implementation of Ramadan Fasting Algorithm for Singaporeans With Type 2 Diabetes
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joyce Lee (Other)
Collaborators: National University of Singapore (Other); Tan Tock Seng Hospital (Other); National Healthcare Group, Singapore (Other Government)
Responsible Party: Sponsor-Investigator, Joyce Lee, Associate Professor, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/00290
Record Dates: First submitted 2017-09-20; First posted 2017-10-19 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Ramadan Fasting; Randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Other): FAST user
  Interventions: Other: FAST
- Control (Other): Standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: FAST — Fasting Algorithm for Singaporeans with Type 2 Diabetes
  Arms: Intervention
Other: Standard of care — Standard of care
  Arms: Control

SUMMARY:
Background: Ramadan fasting is a religious observance carried out by Muslims all over the world. During Ramadan, Muslims abstain from eating, drinking, and smoking during daylight hours. Although Muslims who are ill, including patients with diabetes, are exempted from fasting, many devoted Muslim patients still insist on fasting despite being advised not to by their healthcare providers. Concerns have been raised over how the practice of fasting may affect the metabolic control of Muslim patients with diabetes. Furthermore, it has also been postulated that the act of fasting may increase the risk of hypoglycemia or glucose toxicity. Although practice algorithms and suggestions on the use of glycemic therapies during fasting have been discussed internationally. they are not generalizable as the observances of Ramadan, duration of fasting and the food ingested differ from one country to another.

Aims: This study aims to develop and implement a clinical practice dose-adjustment algorithm dedicated to the care of Singaporean patients with diabetes who fast during Ramadan.

Hypothesis: The use of clinical practice dose-adjustment algorithm can improve both clinical and humanistic outcomes of patients with type 2 diabetes who wish to fast during Ramadan.

Methods: This is a prospective, randomized, interventional study involving patients with type 2 diabetes who wish to fast for at least 10 days during Ramadan. Eligible patient attending a primary care institution or an outpatient specialist clinic of a tertiary institution will be approached to participate in the study. Consented patients will be randomized to either intervention arm or control arm. Patients in the control arm will receive usual care while patients in the intervention arm will be given additional education session on Ramadan fasting related diabetic management advice and an algorithm that was developed by the study team members based on international guidelines, to guide them on self-management during Ramadan. The primary outcomes will be change in HbA1c. Secondary outcomes include change in fasting blood glucose, post prandial blood glucose, medication adherence and humanistic outcomes. The safety outcomes include self reported incidence of major and minor hypoglycemia as well as hyperglycemia during Ramadan month. All outcomes will be measured at baseline, during Ramadan and at 3 month post Ramadan.

Significance: The validation of the algorithm through this study will ensure effective and safe fasting of patients with type 2 diabetes during Ramadan.

ELIGIBILITY:
Inclusion Criteria:

* All Muslim patients over 21 years of age with Type 2 diabetes who plan to fast for at least 10 days during the month of Ramadan

Exclusion Criteria:

* Patients with history of recurrent hypoglycemia
* Patients who are pregnant
* Patients with eGFR<30ml/min 3 months prior to Ramadan
* Patients with HbA1c > 9.5%
* Patients with DM-related admission 1 month prior to Ramadan
* Patients on active short-term corticosteroid treatment
* Patients who are unable to complete the questionnaires

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline Pre-Ramadan (3 months prior to Ramadan), during Ramadan (+ 4 weeks) and post Ramadan (3 months after Ramadan)
  Change in HbA1c during and after Ramadan from baseline

SECONDARY OUTCOMES:
Incidence of minor and major hypoglycemia | During one month of Ramadan
  Incidence of minor hypoglycemia which is defined as signs and symptoms with known precipitating causes such as irregular eating habits, increased daily activity or other attributes that can be modified. Major hypoglycemia is defined as any hypoglycemic symptoms that require the help from another person.
Incidence of hyperglycemia | During one month of Ramadan
  Incidence of hyperglycemia which is defined as signs and symptoms of frequent urination, increased thirst or fruity-smelling breath.
Change in fasting blood glucose (FPG) | Baseline Pre-Ramadan (3 months prior to Ramadan), during Ramadan (+ 4 weeks) and post Ramadan (3 months after Ramadan)
  Change in FPG during and after Ramadan from baseline
Change in post-prandial blood glucose | Baseline Pre-Ramadan (3 months prior to Ramadan), during Ramadan (+ 4 weeks) and post Ramadan (3 months after Ramadan)
  Change in 2 hours post meal during and after Ramadan from baseline
Change in blood pressure | Baseline Pre-Ramadan (3 months prior to Ramadan), during Ramadan (+ 4 weeks) and post Ramadan (3 months after Ramadan)
  Change in BP during and after Ramadan from baseline
Change in lipid panel | Baseline Pre-Ramadan (3 months prior to Ramadan) and post Ramadan (3 months after Ramadan)
  including LDL, TG, TC, HDL
Change in general health status | Baseline Pre-Ramadan (3 months prior to Ramadan) and during Ramadan (+ 4 weeks)
  EQ-5D-5L
Change in diabetes-related distress | Baseline Pre-Ramadan (3 months prior to Ramadan) and during Ramadan (+ 4 weeks)
  Problem Area in Diabetes (PAID)
Change in diabetes-specific quality of life | Baseline Pre-Ramadan (3 months prior to Ramadan) and during Ramadan (+ 4 weeks)
  Audit of Diabetes Dependent Quality of Life (ADDQoL)
Change in diabetes treatment satisfaction | Baseline Pre-Ramadan (3 months prior to Ramadan) and during Ramadan (+ 4 weeks)
  Diabetes Treatment Satisfaction Questionnaires (DTSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Lee, Pharm D, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - Tan Tock Seng Hospital, Singapore
  - National Healthcare Group Polyclinic (Bukit Batok), Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SWH, Chen WS, Sellappans R, Md Sharif SB, Metzendorf MI, Lai NM. Interventions for people with type 2 diabetes mellitus fasting during Ramadan. Cochrane Database Syst Rev. 2023 Jul 12;7(7):CD013178. doi: 10.1002/14651858.CD013178.pub2. PMID 37435938